CLINICAL TRIAL: NCT01465724
Title: Sympathetic Denervation of the Renal Artery for the Treatment of Obesity-related Hypertension and Insulin Resistance
Brief Title: Denervation of the REnal Artery in Metabolic Syndrome
Acronym: DREAMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Michiel Voskuil, MD, PhD, Prinicpal investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-265
Record Dates: First submitted 2011-10-25; First posted 2011-11-07 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Insulin Resistance; Blood Pressure
Keywords: Insulin resistance; Insulin sensitivity; HOMA-IR; blood pressure; Renal denervation; renal sympathetic denervation; renal ablation
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal denervation (Experimental)
  Interventions: Procedure: Renal denervation

INTERVENTIONS:
Procedure: Renal denervation — percutaneous selective renal sympathetic denervation with the use of the Symplicity Catheter system.
  Other Names: Symplicity Catheter system

SUMMARY:
The current prevalence of hypertension as part of the metabolic syndrome is substantial and is increasing with the rise of obesity worldwide. Chronic elevation of sympathetic nervous system (SNS) activity has been identified as a common and key factor in disease states as obesity-related hypertension (ORH). The renal sympathetic nerves are a major contributor to the complex pathophysiology of this elevated SNS activity. Percutaneous renal denervation (PRDN), the deliberate disruption of the nerves connecting the kidneys with the central nervous system, has been shown to be an effective means of modulating elevated SNS activity.

This current study is an observational feasibility study, with the aim to investigate the effect of renal denervation on changes in insulin resistance and blood pressure in patients with obesity related hypertension. The investigators will study different variables: a laboratorial set, a set of blood pressure measurements and a set of investigations in the vascular laboratory.

Hypothesis

* The investigators hypothesize that renal denervation has a beneficial effect on insulin resistance.
* The investigators hypothesize that there will be no complications related to the device or procedure.

DETAILED DESCRIPTION:
Objectives: The objectives of this study are: to compare changes in insulin resistance in patients with ORH after RDN; to evaluate the safety of PRDN in this patient group; to compare changes in blood pressure, laboratory parameters, arterial stiffness and SNS-activity after PRDN.

Study design: Prospective observational feasibility-study.

Study population: Patients with a high fasting glucose (fasting serum glucose ≥5.6 mmol/L(100 mg/dL)) and with an ambulatory systolic blood pressure >130mmHg.

Major endpoints: The effect of RDN on: insulin resistance, blood pressure and major adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a high fasting glucose (fasting serum glucose ≥5.6 mmol/L (≥100 mg/dL)), without the use of antidiabetic drugs at the time of inclusion AND should have a 24 hour ambulatory SBP >130 mmHg, without the use of antihypertensive drugs at the time of inclusion.
* Patients should fulfil one or more other criteria to meet the definition of the metabolic syndrome.
* Individual understands the study procedures, alternative treatments available, risks involved with the study and voluntarily agrees to participate by giving informed consent.
* Individual is over 18 years of age on the day of signing informed consent.

Exclusion Criteria:

* SBP >180 mmHg and/or DBP >110 mmHg during one or more screening measurements.
* 24-hour ambulatory SBP >170 mmHg and/or 24-hour ambulatory DBP >100 mmHg at time of inclusion.
* Individual is treated with more than one type of antihypertensive medication at time of inclusion.
* Individual is treated with more than one type of drug for diabetes mellitus 2 at time of inclusion and/or the medication for DM type 2 can not be stopped.
* Individual has a treatable secondary cause of hypertension.
* Individual has renal artery anatomy that is ineligible for treatment.
* Individual has an estimated glomerular filtration rate (eGFR) of <45mL/min/1.73m2, using the MDRD calculation.
* Individual has type 1 diabetes mellitus.
* Individual has experienced a myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 6 months of the screening visit, or has widespread atherosclerosis, with documented intravascular thrombosis or unstable plaques.
* Individual has scheduled or planned surgery or cardiovascular intervention in the next 6 months.
* Individual has hemodynamically significant valvular heart disease for which reduction of BP would be considered hazardous.
* Individual has an implantable cardioverter defibrillator (ICD) or pacemaker whose settings cannot allow for RF energy delivery.
* Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, haemophilia, or significant anaemia).
* Individual is pregnant, nursing or planning to be pregnant.
* Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
* Individual is currently enrolled in another investigational drug or device trial.
* Individual is currently being treated with any of the following medications:

  * Drugs that cause salt retention (e.g., systemic corticosteroids and fludrocortisone)
  * Acenocoumarol or phenprocoumon that cannot be temporarily stopped for the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Difference in Insulin resistance before and 12 months after renal denervation | T=0, T=6 months, and t=12 months
  To investigate the influence of percutaneous renal sympathetic denervation on insulin resistance. Hereby evaluating an Oral Glucose Tolerance Test before and after renal denervation

SECONDARY OUTCOMES:
Difference in blood pressure before and after renal denervation | t=0, t=6 months, and t=12 months
Safety | one year
  Major adverse events, characterized by myocardial infarction, cerebrovascular accident or all-cause mortality.
Fasting glucose before and after renal denervation | t=0 and t=12 months
Change in Muscle sympathetic nerve activity (MSNA)after renal denervation | t=0 and t=6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Voskuil, MD, PhD, Principal Investigator — UMC Utrecht; Willemien Verloop, MD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands